CLINICAL TRIAL: NCT01765205
Title: The Efficacy of Newborn Screening for Critical Congenital Heart Disease
Brief Title: Newborn Screening for Critical Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 118-2010
Record Dates: First submitted 2012-12-06; First posted 2013-01-10 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Congenital Cardiovascular Malformation
Keywords: congenital cardiovascular malformation; newborn
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Newborns with Pulse oximetry: Up to 50 healthy newborn participants will receive 15 minutes of pulse oximetry to determine the effectiveness of measuring somatic oxygen saturation.
  Interventions: Device: Pulse Oximetry using the INVOS (In Vivo Optical Spectroscopy) Cerebral/Somatic Oximeter
- CHD infant with pulse oximetry: Up to 10 infants diagnosed with congenital heart disease will receive 15 minutes of pulse oximetry using the INVOS Cerebral/Somatic Oximeter to determine the effectiveness of measuring somatic oxygen saturation.
  Interventions: Device: Pulse Oximetry using the INVOS (In Vivo Optical Spectroscopy) Cerebral/Somatic Oximeter

INTERVENTIONS:
Device: Pulse Oximetry using the INVOS (In Vivo Optical Spectroscopy) Cerebral/Somatic Oximeter — Up to 50 healthy infants and up to 10 infants with CHD will receive the pulse oximetry using the INVOS Cerebral/Somatic Oximeter for 15 minutes to determine the effectiveness to measure somatic oxygen saturation. The pulse oximeter will be placed on the infants forehead with a hat and around the infants thigh to measure oxygen saturation.
  Other Names: Healthy Newborns with Pulse oximetry

SUMMARY:
Previous studies have examined the usefulness of pulse oximetry or oxygen saturation to screen for left-sided cardiac lesions. These studies have shown that the occurrence of critical congenital cardiac malformations among asymptomatic newborns is high; the technique of pulse oximetry is reliable for detection of ductal dependant left-sided lesions, simple to operate(requires little time and can be done in the newborn nursery) and is cost effective; there is effective follow-up test (heart ultrasound) and available interventions have an effect on outcome for diagnosed newborns. The importance of this research project is to examine the overall helpfulness of measuring oximetry in newborn infants using somatic oximetry, as well ast to prepare for a population based study in the state of Florida.

DETAILED DESCRIPTION:
This study will evaluate up to 50 unaffected newborns and up to 10 known congenital heart disease (CHD) newborns using a new oximetry system. This system is interfaced to a laptop computer which computes the difference between central and lower extremity peripheral values, upper and lower body peripheral values, and records all data. This information may differentiate unaffected newborns and CHD newborns, and determine the effectiveness of pulse oximetry as a newborn screening for congenital cardiovascular malformations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 12 hours -2 weeks.
* Newborns with identified congenital heart disease or newborns without identified congenital heart disease.
* Congenital Heart Diagnosis: Total Anomolous Pulmonary Venous Return (TAPVR); Atrio-ventricular Septal Defect ( AVSD); Coarctation of the Aorta; Critical Aortic Stenosis; other cyanotic legions including Hypoplastic Left Heart Syndrome ( HLHS)

Exclusion Criteria:

* Have any concurrent condition which, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 12 Hours to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy newborns and newborns diagnosed with congenital cardiovascular malformations
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To measure the oxygen saturation using pulse oximetry. | Baseline
  The oxygen saturation will be measured by pulse oximetry on an infant's skin on the forehead and thigh. These two numbers will be recorded as whole numbers on the machine and will be compared to both groups of infants.

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Byrne, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States